CLINICAL TRIAL: NCT06197126
Title: A Prognostic Model Based on MRI for Cervical Cancer Patients Treated With Radiotherapy
Brief Title: MRI-based Signatures for Survival Prediction in Cervical Cancer With Radiotherapy
Status: Not yet recruiting | Type: Observational
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: SY-GO001
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Cervical Cancer; Radiotherapy; Prognostic Model; MRI
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cervical cancer patients with radiotherapy: Radiotherapy is the main treatment strategy with an overall dose of over 75Gy.
  Interventions: Radiation: Treatment mainly composed of external pelvic beam radiotherapy (EBRT) followed by individualized high-dose-rate intracavitary brachytherapy (HDR-ICBT) .

INTERVENTIONS:
Radiation: Treatment mainly composed of external pelvic beam radiotherapy (EBRT) followed by individualized high-dose-rate intracavitary brachytherapy (HDR-ICBT) . — The chemotherapy regimens included cisplatin (40 mg/m2) or nedaplatin (80 mg/m2) monotherapy or combined with paclitaxel (135 mg/m2) every three weeks during radiotherapy.
  Other Names: concurrent chemothearpy

SUMMARY:
This study aims to validate the value of tumor involvement features based on MRI in cervical cancer, facilitate the development of a more appropriate model for risk stratification, and help patients with varying risk profiles make appropriate decisions in treatment selection and follow-up plans.

DETAILED DESCRIPTION:
Even with the development of advanced technology, the prognosis for CC patients who received radiotherapy is still an intractable problem. Almost 40% suffered disease recurrence among locally advanced patients after radiotherapy and the reported 5-year overall survival is 50-70%. The present FIGO staging is controversial in pre-treatment assessment, which is mainly based on physical examination. An ambiguous diagnosis leads to different treatment strategies and follow-up plans, which is associated with prognosis non-improvement. Incorporation of the tumor involvement features based on the MRI into pre-treatment assessment could standardize and improve the consistency and repeatability of diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* (1) pathologically confirmed CC, (2) initially treated in our center

Exclusion Criteria:

* (1) lack of pre-treatment MRI, (2) prior anti-tumor treatment, (3) pelvic surgery history, (4) incomplete therapy, (5) loss of follow-up

Ages: 20 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cervical cancer patients received definitive radiotherapy with pre-treatment MRI.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival | 1-36 months
  the interval from diagnostic day to death or the last follow-up

SECONDARY OUTCOMES:
progression-free survival | 1-36 months
  the interval from diagnostic day to death, the last follow-up, or the onset of regional recurrence or distant metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Cibula D, Potter R, Planchamp F, Avall-Lundqvist E, Fischerova D, Haie Meder C, Kohler C, Landoni F, Lax S, Lindegaard JC, Mahantshetty U, Mathevet P, McCluggage WG, McCormack M, Naik R, Nout R, Pignata S, Ponce J, Querleu D, Raspagliesi F, Rodolakis A, Tamussino K, Wimberger P, Raspollini MR. The European Society of Gynaecological Oncology/European Society for Radiotherapy and Oncology/European Society of Pathology guidelines for the management of patients with cervical cancer. Radiother Oncol. 2018 Jun;127(3):404-416. doi: 10.1016/j.radonc.2018.03.003. Epub 2018 May 1. PMID 29728273
- [Background] Matsuo K, Shimada M, Nakamura K, Takei Y, Ushijima K, Sumi T, Ohara T, Yahata H, Mikami M, Sugiyama T. Predictors for pathological parametrial invasion in clinical stage IIB cervical cancer. Eur J Surg Oncol. 2019 Aug;45(8):1417-1424. doi: 10.1016/j.ejso.2019.02.019. Epub 2019 Feb 18. PMID 30846298
- [Background] Jiang W, He T, Liu S, Zheng Y, Xiang L, Pei X, Wang Z, Yang H. The PIK3CA E542K and E545K mutations promote glycolysis and proliferation via induction of the beta-catenin/SIRT3 signaling pathway in cervical cancer. J Hematol Oncol. 2018 Dec 14;11(1):139. doi: 10.1186/s13045-018-0674-5. PMID 30547809
- [Background] Lindegaard JC, Petric P, Lindegaard AM, Tanderup K, Fokdal LU. Evaluation of a New Prognostic Tumor Score in Locally Advanced Cervical Cancer Integrating Clinical Examination and Magnetic Resonance Imaging. Int J Radiat Oncol Biol Phys. 2020 Mar 15;106(4):754-763. doi: 10.1016/j.ijrobp.2019.11.031. Epub 2019 Nov 30. PMID 31794837
- [Background] Balcacer P, Shergill A, Litkouhi B. MRI of cervical cancer with a surgical perspective: staging, prognostic implications and pitfalls. Abdom Radiol (NY). 2019 Jul;44(7):2557-2571. doi: 10.1007/s00261-019-01984-7. PMID 30903231
- [Background] Salib MY, Russell JHB, Stewart VR, Sudderuddin SA, Barwick TD, Rockall AG, Bharwani N. 2018 FIGO Staging Classification for Cervical Cancer: Added Benefits of Imaging. Radiographics. 2020 Oct;40(6):1807-1822. doi: 10.1148/rg.2020200013. Epub 2020 Sep 18. PMID 32946322
- [Background] Tsuruoka S, Kataoka M, Hamamoto Y, Tokumasu A, Uwatsu K, Kanzaki H, Takata N, Ishikawa H, Ouchi A, Mochizuki T. Tumor growth patterns on magnetic resonance imaging and treatment outcomes in patients with locally advanced cervical cancer treated with definitive radiotherapy. Int J Clin Oncol. 2019 Sep;24(9):1119-1128. doi: 10.1007/s10147-019-01457-3. Epub 2019 May 11. PMID 31079257
- [Background] Bhatla N, Singhal S, Dhamija E, Mathur S, Natarajan J, Maheshwari A. Implications of the revised cervical cancer FIGO staging system. Indian J Med Res. 2021 Aug;154(2):273-283. doi: 10.4103/ijmr.IJMR_4225_20. PMID 35295012
- [Background] Ren J, Li Y, Yang JJ, Zhao J, Xiang Y, Xia C, Cao Y, Chen B, Guan H, Qi YF, Tang W, Chen K, He YL, Jin ZY, Xue HD. MRI-based radiomics analysis improves preoperative diagnostic performance for the depth of stromal invasion in patients with early stage cervical cancer. Insights Imaging. 2022 Jan 29;13(1):17. doi: 10.1186/s13244-022-01156-0. PMID 35092505